CLINICAL TRIAL: NCT01852838
Title: The Contribution of Induced Glycolysis to the Exhaled Volatile Organic Compounds' (VOCs) Signature in Lung Cancer
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Principal Investigator, Dr. Nir Peled MD, PhD, Head, Thoracic Cancer Research and Detection Center- MD PhD FCCP, Sheba Medical Center
Other Study IDs: SHEBA-12-9716-NP-CTIL
Record Dates: First submitted 2013-04-08; First posted 2013-05-14 (Estimated); Last update posted 2014-02-21 (Estimated); Status verified 2014-02

CONDITIONS: Lung Cancer
Keywords: lung cancer; volatile organic compounds; Warburg effect; early detection
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Lung cancer patients, pre treatment: Patients who have diagnosed with lung cancer before treatment
- High risk patients for lung cancer: high risk patients who are age and co-morbidity matched controls without proof of lung cancer.

SUMMARY:
Lung cancer is the most lethal cancer, killing ~1.3 million people worldwide every year. Early diagnosis could increase its survival by 3-4 folds. Therefore the yield of screening for lung cancer is not a question anymore and the urgent unmet need is to define the group that is under a high risk for lung cancer.

Our lab is focusing on revealing non-invasive biomarkers as for early detection of lung cancer. This study specifically focuses on biomarkers that are found in exhaled breath. These biomarkers are known as volatile organic compounds (VOCs).The VOCs' profile can discriminate between those who suffer from lung cancer and healthy individuals.

It is well established that a cancer cell can activate their glycolysis (glucose degradation) pathway in order to survive. This links malignant processes with this basic biochemical, metabolic cycle. This study will focus on the unique processes incurred by glycolysis in the tumor cells and its effect on the surrounding environment. By better understanding and revealing the exact mechanism, it will become possible to identify the biomarkers released by malignant cells that use glycolysis as a source of energy.

This study's goal is to identify and analyze those distinguishing VOCs. The hope is that these VOCs will provide a new innovative possibility of developing the so desperately needed, early-detection lung cancer screening method.

This research will collect and analyze the exhaled breath of participants. The exhaled breath will be obtained before and after a glucose challenge test, in which the participant is asked to drink a solution containing water and glucose. This study will involve a total of seventy participants, fifty of which currently suffer from active lung cancer, while the remaining participants belong to a high-risk group.

DETAILED DESCRIPTION:
The Contribution of induced Glycolysis to the Exhaled Volatile Organic Compounds' (VOCs) Signature in Lung Cancer

Abstract:

Lung cancer is infamous for its cruel mortality rates as it is the most lethal cancer in both men and women. Unfortunately, most lung cancers are detected and diagnosed at a very advanced stage and this complicates treatment options. Therefore, there is dire, unmet need to develop an effective, highly sensitive, highly specific and non-invasive screening method. The solution to this problem may be found in volatile organic compounds (VOCs) which are organic molecules identified in exhaled breath. These VOCs differ between those individuals who suffer from lung cancer and healthy individuals. Seeing as increased glycolysis is one of the characteristic patterns of malignancies, the purpose of this study is to determine the contribution of induced glycolysis to these exhaled VOCs. Therefore, this study will compare exhaled breath samples in individuals who suffer from lung cancer before and after a glucose challenge test. This study aims to better understand the mechanisms involved in order to identify the distinguishing VOCs. This may aid in developing the so necessary diagnostic means for lung cancer screening.

1. Introduction:

   Lung cancer is the moth lethal cancer in both men and women. [1] There are two main classes of lung cancer: the first, Small Cell Lung Cancer (SCLC) which is often referred to as Oat Cell Cancer, and the second being Non-Small Cell Lung Cancer (NSCLC), which constitutes the majority of cases of lung cancer. [2] Unfortunately, most lung cancer detection and diagnosis is performed when the cancer is in an advanced, metastatic stage in which surgery is not a viable treatment option. [3] Thus, detection and diagnosis its early stages may significantly improve the five year survival rate as well as provide the possibility of a cure.

   An effective, non-invasive lung cancer screening method for distinguishing biological markers found in high-risk groups has yet to be developed. Lately, researchers have begun considering Volatile Organic Compounds' (VOCs) templates as a possible means for early detection. These VOCs can be retrieved and isolated from exhaled breath samples. The VOCs reflect the unique metabolic and biochemical activity in malignant cells. This association has been proven in several researchers as well as in our own group [4] who has shown that not only can VOCs distinguish between healthy and affected individuals, but they can even discern between SCLC and NSCLC. [5, 6] The current research will focus on the detection, identification and the characterization of these unique biological markers found in the exhaled breath of those who suffer from lung cancer. Amongst those VOCs which are detected, this research will specifically focus on those VOCs which hold the potential to be incorporated into an effective, non-invasive screening method for lung cancer.

   Carcinogenesis is a process that is bound to somatic evolution. One of the most popular evolutionary advantages found in malignant, metastatic cells is the increased uptake of glucose through the process of glycolysis. This glycolysis process is unique to malignant cell because it is most pronounced in anaerobic conditions, whereas healthy cells most often perform glycolysis in aerobic conditions. Anaerobic glycolysis- the process of the conversion of glucose to lactic acid in the presence of oxygen- is also known as the "Warburg Effect" after Otto Warburg who discovered this characteristic. [7]

   Thus, some of the distinguishing processes found in malignant cells are the exceeded rate of substance exchange and increased glucose degradation (Warburg Effect). These processes release organic compounds, some of which are released into exhaled breath. Therefore, this research will examine the relationship between a glucose challenge test and its effect on the pattern on VOCs in exhaled breath.
2. Research Goals:

   The template for organic particles in exhaled breath discriminates between those individuals who suffer from active lung cancer from those individuals who are considered healthy. The purpose of this study is to examine the contribution of the process of glycolysis to this unique template. Being that the process of glycolysis is accelerated in malignant cells, we hypothesize that the glucose challenge test will express VOC in those individuals who suffer from the disease. These findings can contribute to the development of diagnostic tools for lung cancer.
3. Hypothesis:

   We hypothesize that the Warburg Effect is an essential component in the creation of VOCs that are unique to lung cancer, and therefore, that the glucose challenge test will increase the production of these VOCs. These markers hold the potential to create a more effective, non-invasive screening method with improved sensitivity and specificity.
4. Methods:

4.1 Research Design: This research is an observational case-control study assesses the comparison between the VOCs samples obtained from exhaled breath samples and blood tests taken before and after a glucose challenge test. The glucose challenge test involves drinking a solution which contains 75 grams of glucose and a waiting period of 90 minutes between the collection of exhaled breath and blood samples. There is a need to fast for six hours before this test. In addition, a clinical assessment will be performed based on the medical anamnesis and on existing, current medical information.

4.2 Study Population: The goal of this research is to determine if the process of glycolysis contributes to the unique VOC pattern in the exhaled breath of those who are affected with lung cancer. The participants will be chosen from individuals that are currently being treated in pulmonology clinics for various reasons. The control group will include participants that have been identified as high-risk individuals for lung cancer, whereas the study group will include participants who suffer from active lung cancer but have not yet begun any form of medical treatment.

The recruitment process will be performed in two consecutive stages. In the first stage, twenty patients from the study group will be compared to the twenty participants from the control group. At this point, a preliminary assessment of the data will be performed to find differences in the VOCs between these two groups. Only in the event that these differences are found will the research go on to the second stage, in which 30 more participants will be recruited and tested for the study group.

The control group as previously mentioned will include 20 participants that do not have lung cancer, but are similar to the research group in terms of age, gender, medical history, and history of smoking. This classification will be performed based off the self-report surveys completed by the participants.

Exclusion criterions for the study population are as follows:

1. Patients that are uninterested to participant and/or unable to sign a consent form
2. Lung Cancer patients who have begun treatment prior to this research
3. Patients who are unable to complete this research and/or the follow up visits
4. Individuals that suffer from diabetes

4.3 Research Variables:

The main variables which will be used to test our hypothesis are as follows:

* Epidemiological variables of the participants
* Quantitative data defining the malignant cells ( TMN, the size of the tumor, number of metastases and their location)
* The glucose levels( via a dipstick) before and after the glucose challenge test (requires a fast of 6 hours prior to the test)
* The VOCs pattern obtained from the exhaled breath samples and the characterization of these molecules via the GCMS method.

4.4 Research Methods:

Medical Anamnesis:

A collection of the details of the patient's medical history will be obtained. Information such as gender, age, medical history, consumption of tobacco and family history will be noted. In addition, information which quantifies and qualifies the malignant cells (if present) will be collected and recorded. This includes details such as the type of tumor as well as its place, volume, histological characteristics and imaging results. Some of the medical information will be obtained from pre-existing updated medical records.

Exhaled Breath Test:

Each participant will undergo an exhaled breath test before and after the glucose challenge test with a lay period of 90 minutes in between the tests.

The detailed explanation regarding the process of collection of the exhaled breath samples:

The patient will exhale 3 breaths (with 750 ml in each exhaled breath) into appropriate Mylar bags in a sterile area with technology that ensures that the exhaled breath is isolated and unaffected from the external environment. The contents of the Mylar bags will be stored in TENAX samples which preserves the samples for a period of six months. The samples will undergo additional analysis at the Israel Institute of Technology (Technion) under the auspices of Professor Haim Hussam. Each sample will be analyzed for the purposes of identifying VOCs via the GC-MS method. The sample will undergo additional processing such as SPME (pre-concentration into solid-phase micro extraction). The SPME will be transferred to the GC-MS. The GC-MS method allows for the identification of the compounds in a short period of time via the use of chromatographic and spectroscopic instruments. The spectroscopic instrument will undergo additional analysis via the AOS instrument. The AOS includes detectors which are conjugated to nano-particles of gold. Each detector identifies a wide variety of VOCs in accordance to their location and concentration which cause varying levels of resistance. This response is recorded and will undergo statistical analysis via PCA to focus on the specific VOC patterns found in the sample.

The detailed explanation of the process of the glucose challenge test is as follows:

The participant is requested to drink a sugary solution (273 ml) constituted from 75 grams of glucose and water. The test requires that the participant fast for a period of 6 hours before the test. After drinking the solution, the participant must wait a lay period of 90 minutes before the retest of his or her exhaled breath. In addition, the level of glucose will be tested by a dipstick before drinking the solution, and after the 90 minute lay period.

4.5 Statistical Analysis: The sample size is 70 persons ( 40 persons in the first stage, and an additional 30 participants in the second stage as explained above).

The expectation is that there will be a significant difference between the VOC template before and after the glucose challenge test. The estimated difference of effect is around 30%, with the assumption that the sampling error stands at around 10% and with a confidence interval of 95%. The number of necessary participants needed in order to achieve results with statistical significance and size effect ranges from approximately 20-25 persons.

The information from the AOS which recorded the changes in resistance will be analyzed via PCA to focus on the specific VOC pattern changes obtained in each sample.

The remaining variables which were measured quantitatively will be presented in averages with their corresponding standard deviations. Those variables that were obtained quantitatively will be presented as percentages.

Statistical analysis for significance will be performed by the following statistical tests: Student's T Test, Chi-Square, Analysis of Variance (ANOVA), and the Kruskal-Wallis test. All statistical tests will be performed on the SPSS computer program.

ELIGIBILITY:
Inclusion Criteria:

* 50 individuals who currently suffer from lung cancer, who have not yet begun any medical treatment
* 20 individuals who have been defined as high-risk patients for lung cancer by the Research and Detection Unit for Thoracic malignancies at the Sheba Medical Center, Tel Hashomer, Israel

Exclusion Criteria:

* individuals who suffer from diabetes
* Individuals who suffer from lung cancer, and are currently being treated
* minors ( under the age of 18)

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The population will include a total of 70 participants, 50 of which currently suffer from lung cancer, and have not yet begun any form of medical treatment whilst the remaining group consists of 20 individuals who have been defined as high-risk patients for lung cancer by the Research and Detection Unit for Thoracic malignancies at the Sheba Medical Center, Tel Hashomer, Israel.
Sampling Method: Non-Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2013-09; Primary Completion 2015-04 (Estimated); Study Completion 2015-04 (Estimated)

PRIMARY OUTCOMES:
Diagnostic VOC signature for lung cancer | 2 year
  Each breath sample will be analyzed to identify VOCs via the GC-MS and Artificaial olfactory System AOS. We expect a significant difference between the VOC template before and after the glucose challenge test. The estimated difference of effect ~ 30%, with a sampling error ~ 10% and CI ~ 95% and sample size of 20-25 persons.
  The information from the AOS which recorded the changes in resistance will be analyzed via PCA to focus on the specific VOC pattern changes obtained in each sample.
  The remaining variables which were measured quantitatively will be presented in averages with their corresponding standard deviations. Those variables that were obtained quantitatively will be presented as percentages.
  Statistical analysis for significance will be performed by the following statistical tests: Student's T Test, Chi-Square, Analysis of Variance (ANOVA), and the Kruskal-Wallis test.

CONTACTS AND LOCATIONS:
Overall Officials: Nir Peled, MD PhD FCCP, Principal Investigator — Sheba Medical Center
Locations (1):
- Sheba Medical Center, Ramat Gan, Ramat Gan, Israel